CLINICAL TRIAL: NCT05512871
Title: A Mobile Health (mHealth)-Enabled Lifestyle Intervention Among Women With History of Gestational Diabetes (GDM): a Pilot Randomized Controlled Trial
Brief Title: A Mobile Health-enabled Lifestyle Intervention Among Women With History of Gestational Diabetes(GDM)
Acronym: Reverse-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: National University Polyclinics, Singapore (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Johan Eriksson, Executive Director & Programme Director (Human Development), Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/00843
Record Dates: First submitted 2022-07-25; First posted 2022-08-23 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Gestational Diabetes Mellitus in Pregnancy; Diabetes, Gestational
Keywords: Healthy women, Gestational Diabetes Mellitus history, GDM history, mobile health apps
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The study is a parallel 2-arm, single-centre randomized controlled trial based on 1:1 allocation ratio:
  Group1 (Intervention group) - Oura ring with Oura App + HealthifySG App (receive lifestyle interventions via HealthifySG App) Group 2 (Control group) - Oura ring with Oura App alone (without lifestyle interventions)
Masking Description: 60-80 female subjects will be randomized to either Group 1 (Intervention group) or Group 2 (Control group) based on 1:1 allocation. HealthifySG App will only be installed on the phones of subjects for Group 1(Intervention group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Intervention group) (Experimental): Group 1 (Intervention group) :Oura ring with Oura App + HealthifySG App (receive lifestyle interventions via HealthifySG App)
  Interventions: Behavioral: Personalized mHealth intervention to promote short-term metabolic and mental health among women with a history of Gestational Diabetes Mellitus (GDM)
- Group 2 (Control group) (Other): Group 2 (Control group) : Oura ring with Oura App alone (without lifestyle interventions)
  Interventions: Behavioral: Personalized mHealth intervention to promote short-term metabolic and mental health among women with a history of Gestational Diabetes Mellitus (GDM)

INTERVENTIONS:
Behavioral: Personalized mHealth intervention to promote short-term metabolic and mental health among women with a history of Gestational Diabetes Mellitus (GDM) — The study aim to conduct lifestyle intervention trials to examine the feasibility, efficacy, and cost-effectiveness of the mHealth approach in preventing them from developing Type 2 Diabetes in the future. This pilot study will primarily aim to determine the feasibility of our intervention approaches as well as enhance health literacy and promote healthy lifestyle in the study participants. In the longer term, we hope that the proposed mHealth intervention can be translated to include women from the community setting and involve wider healthcare setting to come together and reduce the burden of Type 2 Diabetes in Singapore.

SUMMARY:
This study aims to explore: (1) the relationship between lifestyle factors (eating, movement behaviour, sleep and stress) and glycaemic profile, and (2) the feasibility of delivering lifestyle intervention through the proposed mHealth strategy.

DETAILED DESCRIPTION:
A 2-week observational period, followed by a 8-week parallel 2-arm, single-centre, randomized controlled trial (RCT) study involving 60-80 multi-ethnic healthy women (Chinese, Malay, Indian, others) subjects aged between 21 and 45 years who had a previous diagnosis of Gestational diabetes mellitus (GDM).

Type 2 diabetes is the most common type of diabetes and if left untreated or is ill-managed, can lead to detrimental long-term health problems such as heart disease, kidney disease and stroke. Type 2 diabetes is often related to lifestyle and develops over time; with proper interventions, it could be avoided in some cases. GDM stands for Gestational Diabetes Mellitus and can occur in some pregnant women, usually from week 24 of pregnancy. Women with a history of GDM have also been connected to a lifetime risk of developing type 2 diabetes and cardiovascular disease. In Singapore, it is estimated that 4 in 10 women with GDM could develop pre-diabetes or diabetes within five years of their pregnancy. Therefore, postpartum follow-up is essential in early detection of, preventing or delaying the development of Type 2 diabetes in this group.

The study hypothesize that there is an association between glycaemic profile and daily lifestyle (i.e. eating behavior, physical activity sleep and stress) among women with a history of GDM. The study also hypothesize that it is feasible to adopt a holistic approach and introduce a personalized mHealth intervention to promote metabolic and mental health among women with a history of GDM. The study is a parallel 2-arm, single-centre randomized controlled trial based on 1:1 allocation ratio.

The study arms are; Group 1 (Intervention group) and Group 2 (Control group). The study will begin with baseline data collection (anthropometric measures, body composition, biochemistry tests, questionnaires) and 14-day observation of interstitial glucose and lifestyle (diet, physical activity, sleep and stress). Every subject, irrespective of their group allocation, will use Oura ring and Oura App throughout the study duration. Every subject randomized to Group 1( Intervention group) will additionally receive HealthifySG App which provides personalized lifestyle interventions that last for 4 weeks. Lifestyle recommendations (targeting diet, physical activity, sleep and stress) will be delivered by study team member through the HealthifySG App on a weekly basis. On the contrary, subjects randomized to Group 2 (Control group) will not receive the HealthifySGApp and lifestyle interventions during this period. Subsequently, both groups will be followed-up for 4 weeks.

The overall aim of the REVERSE DIABETES programme is three pronged: (1) to be more proactive in screening to identify women with a history of GDM in polyclinics and the community, (2) to explore the potential of mobile health (mHealth) strategies to engage these women and deliver holistic and personalized interventions for promoting metabolic health and mental wellbeing, and (3) to engage primary care physicians to use mHealth if proven acceptable and useful in the long term follow up of these GDM women in the polyclinics and communities. We hope to optimize the preventive measures within the community in the long term.

Based on the above considerations, conducting a pilot randomized controlled trial would allow the study team to: (1) better understand the women's lifestyle behaviours and preferences, (2) validate the devices used for measuring lifestyle behaviours, (3) examine the feasibility of the proposed mHealth intervention and personalized lifestyle recommendation, (4) evaluate the initial effects and cost-effectiveness of the intervention, and (5) identify other benefits and potential risk of the proposed idea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers (age 21-45 years)
* A history of GDM in the past 5 years
* Not planning to conceive during the study period
* Not performing full breastfeeding during the study period
* Own a smart phone(mobile phone) compatible with study App (Android v10 and above)
* Proficient in English language
* Plan to stay in Singapore for the next 1 year
* Willing to comply to study protocol
* Able to provide a written informed consent

Exclusion Criteria:

* Current and/or previous diagnosis of diabetes except GDM
* Currently pregnant
* Given birth within last 12 weeks
* Following special diet or dietary restriction
* Experiencing severely limited mobility (e.g. wheelchair bound, need walking aid etc.)
* Diagnosed with malnutrition, eating disorder, severe insomnia
* Diagnosed with cancers, unstable heart related diseases, severe kidney disease
* Diagnosed with severe unstable mental conditions, dementia or cognitive impairment
* Alcohol or drug abuse
* Medications known to influence glucose metabolism e.g. peroral corticosteroids

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women volunteers who has given birth previously and with a history of GDM within the last 5 years (Post partum 13 weeks and beyond).
Enrollment: 61 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Mobile health application feasibility | 10 weeks
  Number of participants that show a change in lifestyle behaviour through the mobile health application usage.

SECONDARY OUTCOMES:
Oral glucose tolerance test (OGTT) measurements | Week -1 and 10
  Glucose metabolism is measured during baseline visit via a fasting blood test and endpoint visit via the Oral glucose tolerance test (OGTT) blood test. The difference in the blood glucose profile between the baseline and the endpoint visit will determine the effects of the proposed mobile Health intervention.
Change in sleep quality as assessed by the Oura Ring Sleep Score. | 10 weeks
  Participants will be issued a wearable device (Oura ring) to capture durations of deep sleep, rapid eye movement (REM) sleep, light sleep and nightly heart rate. Sleep Score ranges from 0-100, where a higher score reflects better sleep outcome.
Change in daily physical activity levels as assessed by the Oura Ring Activity Score. | 10 weeks
  Participants will be issues a wearable device (Oura ring) to capture durations of activity, inactivity and rest. Activity score ranges from 0-100, where a higher score reflects better balance between activity and rest.
Postprandial glucose | 14 days
  Glucose measurements taken using the Continuous Glucose Monitoring System.
Change in quality of life | Week -1 and 10
  Assessed by the 36-item short form survey (SF-36)
Change in anxiety (if any) | Week -1 and 10
  Assessed by State-Trait Anxiety Inventory (STAI)
Change in depression (if any) | Week -1 and 10
  Assessed by Beck Depression Inventory-II (BDI-II).
Change in intake of meals | 14 days
  Assessed by Electronic diary(E-Diary) by recording the pictures of food items for meals

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Centre (Hdrc), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liew SJ, Soon CS, Chooi YC, Tint MT, Eriksson JG. A holistic approach to preventing type 2 diabetes in Asian women with a history of gestational diabetes mellitus: a feasibility study and pilot randomized controlled trial. Front Clin Diabetes Healthc. 2023 Sep 28;4:1251411. doi: 10.3389/fcdhc.2023.1251411. eCollection 2023. PMID 37841647